CLINICAL TRIAL: NCT05264688
Title: The Role of Novel PET Molecular Imaging Targeting Fibroblast Activation Protein in the Diagnosis of Hepatobiliary Malignancies
Brief Title: The Function of PET Molecular Imaging Targeting Fibroblast Activation Protein in the Hepatobiliary Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yufeng Yuan, professor, Zhongnan Hospital
Other Study IDs: 20220207
Record Dates: First submitted 2022-02-07; First posted 2022-03-03 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hepatobiliary Diseases
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-04 imaging agent — 1.85-3.7 MBq/kg body weight (0.05-0.1 mCi/kg) intravenously

SUMMARY:
Patients with high clinical suspicion of hepatobiliary malignancies should undergo PET/CT examination with two imaging agents, 68Ga-FAPI (fibroblast activation protein inhibitor) and 18F-FDG within one week, and collect tumor tissue. Finally, the PET/CT results were compared with the pathology report to evaluate the role of 68Ga-FAPI PET/CT imaging in the diagnosis of hepatobiliary malignancies

DETAILED DESCRIPTION:
Patients with high clinical suspicion of hepatobiliary malignancies should undergo PET/CT examination with two imaging agents, 68Ga-FAPI (fibroblast activation protein inhibitor) and 18F-FDG within one week. After comprehensive clinical evaluation, if the patient can be treated with surgery, surgery will be performed, and the patient's pathological specimens will be collected after surgery ; If the patient has no possibility of surgery, ultrasound-guided needle biopsy is performed, and biopsy specimens are collected. Finally, the PET/CT results were compared with the pathology report to evaluate the application value of 68Ga-FAPI PET/CT imaging in the diagnosis and staging of hepatobiliary malignant tumors, and to analyze the guiding significance for the treatment decision of hepatobiliary malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign a written informed consent;
2. 18-80 years old (inclusive) male or female;
3. Patients with high clinical suspicion of hepatobiliary malignancy in combination with medical history and imaging studies, etc.
4. Those who obtained pathological diagnosis results through needle biopsy or surgical resection;
5. Have willingness and ability to participate in all research procedures.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. Those who are known to be allergic to the imaging agent 68Ga-FAPI or its excipients;
3. Those who have a history of other malignant tumors in the past;
4. Before the injection of 18F-FDG, the fasting blood glucose level exceeds 11.0mmol/L;
5. Patients with claustrophobia;
6. Those who cannot tolerate lying down for 15-30 minutes;
7. The researchers believe that it is not suitable to participate in this clinical trial;
8. Those who have participated in clinical trials or are participating in other clinical trials within the past month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high clinical suspicion of hepatobiliary malignancies and meeting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
diagnose accordance rate | 2022.1.20-2022.7.30
  Proportion of PET/CT diagnostic reports consistent with pathological results

SECONDARY OUTCOMES:
Standardized Uptake Mean (SUVmean) | 2022.1.20-2022.7.30
  The average of the standard uptake value
Standardized Uptake Maximum (SUVmax) | 2022.1.20-2022.7.30
  The maximum value of the standard uptake value
Tumor Background Ratio | 2022.1.20-2022.7.30
  The ratio of the radiation concentration in the tumor area to the surrounding background
Tumor Metabolic Volume (MTV) | 2022.1.20-2022.7.30
  The metabolically active volume of tumor tissue
Total Glycolysis (TLG) | 2022.1.20-2022.7.30
  Tumor metabolic volume is multiplied by the mean of standard uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided